CLINICAL TRIAL: NCT01116115
Title: The Effects of Dietary Palmitic Acid Triacylglyceride Position on Intestinal Parameters, Anthropometric Parameters and Stool Characteristics in Term Infants
Brief Title: The Effects of Dietary Palmitic Acid Triacylglyceride Position on Intestinal Parameters in Infants (InFat_005)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Fabiana Bar-Yoseph, Enzymotec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: InFat_005
Record Dates: First submitted 2010-04-07; First posted 2010-05-04 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Health Behavior; Disorder of Growth and Development
Keywords: Term Infants; Intestine flora; Stool characteristics
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard vegetable oil based formula (Active Comparator)
  Interventions: Other: Standard vegetable oil based infant formula
- InFat™ based infant formula (Active Comparator)
  Interventions: Other: InFat™ based infant formula
- Breast-fed (No Intervention)

INTERVENTIONS:
Other: InFat™ based infant formula — High sn-2 palmitic acid oil based infant formula
  Other Names: High sn-2 palmitic acid; structured triglyceride
  Arms: InFat™ based infant formula
Other: Standard vegetable oil based infant formula — Standard vegetable oil based infant formula
  Other Names: Standard vegetable oil
  Arms: Standard vegetable oil based formula

SUMMARY:
The purpose of this study is to determine the effect of high sn-2 palmitic acid based infant formula on intestinal parameters in term formula fed infants.

DETAILED DESCRIPTION:
InFatTM is an advanced basic-fat ingredient, which mimics the fat composition and properties of human milk fat and enabling optimal intake of the essential calcium and energy (in the form of fatty acids) and easy digestion. These benefits are the result of a unique fatty acid composition on the glycerol backbone, which ensures high level of palmitic acid at the middle (sn-2) position.

The purpose of this study is to determine the effect of high sn-2 palmitic acid based infant formula on intestinal parameters, anthropometric parameters and stool characteristics in formula fed term infants.

ELIGIBILITY:
Inclusion Criteria:

1. Parental/ legal guardian written inform consent
2. The mother had unequivocally decided not to breast-feed (in formula groups) or the mother had decided to breast feed (in human breast milk group).
3. Term infants of born at 37-42 gestation weeks as determined by menstrual history and corroborated by prenatal US and/or physical examination.
4. Birth weight appropriate for gestational age (AGA).
5. The infant is apparently healthy at birth and entry to study.
6. Apgar after 5 minutes >7
7. Enrolled within their first 7 days of life
8. The infant is a product of normal pregnancy and delivery, including C-section.
9. Parental ability to attend visits and interviews and willing to fill questionnaires.

Exclusion Criteria:

1. Mother health condition: (psychological or physical) or socioeconomic problems that may interfere with the mother's ability to take care of her infant or according to PI discretion may interfere with study results.
2. The infant suffers from a major congenital abnormality, a disease or chromosomal disorder with a clinical significance that can be detected at or around birth.
3. The infant suffers/ed from a disease requiring mechanical ventilation or medication treatment at the first week after birth.
4. The infant suffers from any suspected or known metabolic or physical limitations interfering with feeding or normal metabolism (require a special formula).
5. The infant or mother was treated with antibiotics around birth.

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Intestinal flora composition | Baseline, 5 weeks
  infant feces microbial analysis

SECONDARY OUTCOMES:
Anthropometric measurements | Baseline, 5 weeks
  Body length, weight, and head circumferences
General Health and Well being | Baseline, 5 weeks
  Physical examinations, Health (dieases, doctor visits) and well being (sleeping, crying) questionnaires, medications report

CONTACTS AND LOCATIONS:
Overall Officials: Arie Riskin, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical center, Haifa, Israel

REFERENCES:
- [Derived] Yaron S, Shachar D, Abramas L, Riskin A, Bader D, Litmanovitz I, Bar-Yoseph F, Cohen T, Levi L, Lifshitz Y, Shamir R, Shaoul R. Effect of high beta-palmitate content in infant formula on the intestinal microbiota of term infants. J Pediatr Gastroenterol Nutr. 2013 Apr;56(4):376-81. doi: 10.1097/MPG.0b013e31827e1ee2. PMID 23201699